CLINICAL TRIAL: NCT02591485
Title: Prevention of Post Traumatic Stress Disorder Following Trauma by Attention Control Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yair Bar-Haim (Other)
Responsible Party: Sponsor-Investigator, Yair Bar-Haim, Professor Yair Bar-Haim, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: TASMC - 15 - PH - 0409 - CTIL
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: PTSD
Keywords: PTSD prevention; Acute stress disorder; Attention training; Cognitive bias modification
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Control Training (Experimental): Computerized attention modification training, comprised of six sessions that delivered by internet, in purpose of modulate biases in attention for threat stimuli.
  Interventions: Behavioral: Attention Control Training
- Follow-up only (No Intervention): In this condition, a follow-up interviews will be conducted 3 months since the traumatic event had occurred.

INTERVENTIONS:
Behavioral: Attention Control Training — In the ACT, participants perform six computerized attention training sessions, 10 minutes per training session over six weeks. In each session the dot-probe task is administered. This task is consisted of 160 trials. Each trial began with a centrally-presented fixation cross that then replaced by a pair of words presented. Following that, a target probe appeared in the location previously occupied by one of the words, and participants are requested to discriminate the probe type via button press. Targets appear with equal probability at the location of threat and neutral stimuli, in order to modify the fluctuations in attention allocation.
  Arms: Attention Control Training

SUMMARY:
The purpose of this study is to explore the efficacy of Attention Control Training in preventing the development of Post Traumatic Stress Disorder (PTSD), during the period near after a traumatic event and before PTSD is develop.

Individuals who underwent a traumatic event in the past two weeks will be randomly assigned to either Attention Control Training (ACT), designed to normalize threat-related attention biases or a control conditions: without intervention at all.

Outcome measures will be a diagnosed of PTSD and the level of severity of symptoms derived from the Clinician Administered PTSD Scale (CAPS-5), after 3 month since the traumatic event had occurred.

The investigators expected to find lower ratios of PTSD symptoms in the ACT condition relative to the control condition in which no symptomatic relief is expected.

DETAILED DESCRIPTION:
Background 13-21% out of the people exposed to a potentially traumatic event suffer from Acute Stress Disorder (ASD; American Psychiatric Association, 2013). Findings show that 70% of the people who are diagnosed with ASD during the first month following the traumatic event go on to develop Post-Traumatic Stress Disorder (PTSD; Harvey & Bryant, 1998). PTSD is characterized by re-experiencing of the traumatic event, avoiding situations that remind the event, hypervigilance, and negative feelings and beliefs about the self.

A neurocognitive mechanism that may become disarrayed in PTSD is the threat monitoring system. This system is responsible for monitoring potential threats and for generating adequate behavioral and emotional responses to an ever-changing environment. Recent studies have shown that this system is impaired in PTSD (Iacoviello, et al., 2014; Naim, et al., 2015) and that Attention Control Training (ACT), which balances the system's activity, is related to improvement in PTSD symptoms (Badura-Brack, et al., 2015). Therefore, the aim of the current study is to explore the efficacy of the ACT in preventing the development of PTSD during the period near after the traumatic event and before PTSD is developed.

To this end, the investigators will recruit participants that arrived at the emergency department at the Tel Aviv Sourasky Medical Center ('Ichilov') and experienced a potentially traumatic event (according to the criteria of the Diagnostic and Statistical Manual of mental disorders (the DSM-V). Potential participants will be explained about the study and be asked to provide informed consent to participate. Those who agree to participate will be contacted via a telephone call 10-14 days after the event, and a diagnostic interview will be conducted to determine the presence of ASD, and to determine whether the potential participants meet the inclusion criteria for the study. Those who will exhibit a high level of ASD symptoms will be included in the study.

Those included will be randomly assigned to one of two conditions detailed below. the investigators expected to recruit 4000 candidates at the emergency room, with the expectation that 10% of them (~600 participants) will have ASD 10-14 days later.

Procedure The participants will be individuals who were recently exposed to a potentially traumatic event and arrived at the emergency department in the Tel Aviv Sourasky Medical Center (Ichilov). The study procedure and its aims will be explained to the candidates and they will have to provide written informed consent to be included. The recruitment will be conducted by the research team that will be trained for that purpose and will stay in shifts in the emergency department in coordination with the medical team.

Ten to fourteen days after the event, the participants who agreed to participate and signed the informed consent will be contacted by telephone. In this conversation, a diagnostic interview for ASD (Acute Stress Disorder Interview, ASDI; Bryant, Harvey, Dang, & Sackville, 1998) will be conducted in addition to questions about potential exclusion criteria. Those who demonstrate a high level of ASD symptoms (scores 7 and above in the ASDI), will be randomly assigned to one of two conditions: attention control training (ACT) intervention, or a control condition without intervention.

In the ACT intervention, participants will perform six computerized attention training sessions, 10 minutes per training session over six weeks (a session once a week). Training will be done through a username and password protected website designated for this purpose, so the participants could complete the training from home. In addition, the participants assigned to the control condition without intervention will be followed-up three months after recruitment.

At the end of the intervention period, a clinical interview will be conducted through telephone where a PTSD diagnosis (CAPS-5 interview; Weathers, Blake, Schnurr, Kaloupek, Marx, & Keane ,2013) and other clinical symptoms will be assessed. The interview will be delivered by graduate-level clinical psychology students trained by a senior clinical psychologist. Participants from the control intervention group who will have PTSD in the diagnostic point will be offered to participate in the condition that has shown the most effective improvement.

The duration of the study procedure for each participant will be three months.

ELIGIBILITY:
Inclusion Criteria:

1. The occurrence of a traumatic event (criteria A of PTSD from the DSM-5) in the period of less than a month from the beginning of the study.
2. An ASD diagnosis (score 7 and above in the ASDI).

Exclusion Criteria:

1. A previous traumatic event in the period of three month or less before the current event.
2. Chronic PTSD.
3. A diagnosis of psychotic or bipolar disorders.
4. A diagnosis of a neurological disorder (i.e., epilepsy, brain injury).
5. Suicidal ideation.
6. Drugs or alcohol abuse.
7. Another psychotherapeutic treatment.
8. A pharmacological treatment that is not stabilized in the past 6 months (A stable pharmacological treatment will not be a reason for exclusion from the study).
9. Poor judgment capacity (i.e., special populations).
10. Pregnant women.

Within Study exclusion criteria:

Disagreement to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
A diagnosis of PTSD and a total score of severity symptoms, as driven from the CAPS-5 interview. | 40 minutes
  The Clinician Administered PTSD Scale (CAPS-5), is a structured interview that will be used to make a diagnosis of PTSD according to the DSM-V criteria. This interview is consists of 30 items regarding the frequency and intensity of PTSD symptoms and a total score of severity is been rated (Weathers, Blake, Schnurr, Kaloupek, Marx, & Keane, 2013).

OTHER OUTCOMES:
Total score of the PTSD Checklist (PCL-5). | 10 minutes
  The PCL-5, is a 20-item National Center for PTSD Checklist of the Department of Veterans Affairs. Scores can range from 0 to 80, with higher scores reflecting more symptoms of PTSD (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013).
Total score of depression (PHQ-9). | 10 minutes
  The PHQ-9, is a 10-item scale assess the severity level of depression symptoms.
The Sheehan Disabilities Scale(SDS) | 5 minutes
  The SDS is a functioning impairment rating scale in the domains of work, social, and family life. It contains 3 self-reported items, ranging on severity from 0 to 10 on a 10-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, Prof., Study Director — Tel Aviv University
Locations (1):
- Tel-Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weathers, F., Blake, D., Schnurr, P., Kaloupek, D., Marx, B., & Keane, T., The clinician-administered PTSD scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD at www. ptsd. va. gov, 2013.
- [Background] Weathers, F., B. Litz, T. Keane, P. Palmieri, B. Marx, & P. Schnurr, The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www. ptsd. va. gov, 2013.
- [Background] American Psychiatric Association, Diagnostic and Statistical Manual of Mental Disorders (DSM-5). 2013: American Psychiatric Pub.
- [Background] Harvey AG, Bryant RA. The relationship between acute stress disorder and posttraumatic stress disorder: a prospective evaluation of motor vehicle accident survivors. J Consult Clin Psychol. 1998 Jun;66(3):507-12. doi: 10.1037//0022-006x.66.3.507. PMID 9642889
- [Background] Iacoviello BM, Wu G, Abend R, Murrough JW, Feder A, Fruchter E, Levinstein Y, Wald I, Bailey CR, Pine DS, Neumeister A, Bar-Haim Y, Charney DS. Attention bias variability and symptoms of posttraumatic stress disorder. J Trauma Stress. 2014 Apr;27(2):232-239. doi: 10.1002/jts.21899. Epub 2014 Mar 6. PMID 24604631
- [Background] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075
- [Background] Naim R, Abend R, Wald I, Eldar S, Levi O, Fruchter E, Ginat K, Halpern P, Sipos ML, Adler AB, Bliese PD, Quartana PJ, Pine DS, Bar-Haim Y. Threat-Related Attention Bias Variability and Posttraumatic Stress. Am J Psychiatry. 2015 Dec;172(12):1242-50. doi: 10.1176/appi.ajp.2015.14121579. Epub 2015 Jul 24. PMID 26206076
- [Background] Bryant, R. A., Harvey, A., G., Dang, S., T., & Sackville, T., Assessing acute stress disorder: Psychometric properties of a structured clinical interview. Psychological Assessment, 1998. 10(3): p. 215.